CLINICAL TRIAL: NCT05708859
Title: Effect of Tirzepatide on Progression of Coronary Atherosclerosis Using MDCT
Acronym: T-PLAQUE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Matthew J. Budoff (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 22915-01
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type II Diabetes; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: Double blind Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Active Comparator): Tirzepatide 15mg Prefilled pen for weekly subcutaneous injection over 52 weeks
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo Prefilled pen (volume matched) for weekly subcutaneous injection over 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide 15mg Subcutaneous Solution
  Other Names: Mounjaro
  Arms: Tirzepatide
Drug: Placebo — Volume matched Subcutaneous Solution
  Arms: Placebo

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled, parallel-group phase IV Study evaluating the effects of tirzepatide on atherosclerotic plaque progression assessed by coronary computed tomography angiography (CCTA) in participants with a diagnosis of type II Diabetes (T2DM) and atherosclerosis.

DETAILED DESCRIPTION:
This is a multi-center study in which 120 male and female participants who meet the eligibility criteria will be randomized. Study will assess changes in coronary atheroma volume comparing tirzepatide 15 mg/week plus Standard of Care (SOC), as compared to placebo plus SOC. Potential eligible participants may be prescreened for eligibility prior to the screening visit and must have a diagnosis of atherosclerosis (as assessed by >10% atheroma on CCTA) and T2DM.

Patients must be on a stable medical regiment (>4 weeks on statin therapy and diabetes medications) and undergo screening CCTA to demonstrate coronary plaque. Participant eligibility will be assessed by the Imaging Core Lab.

If the participant meets all entry criteria during baseline visit, then consenting participants will be randomized 1:1 to receive tirzepatide on top of standard of care for treatment period of 12 months. Participants will be asked to maintain stable doses of statins and diabetes medications. Persistent hyperglycemia will be treated by primary physician or endocrinologist,

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 40 years to 80 years of age at signing of informed consent
2. Type 2 DM of minimum 5 years duration with HbA1c ≥7.0% to ≤10.5%
3. Body mass index (BMI) ≥25 kilograms per meter squared (kg/m²)
4. Presence of two discrete coronary artery plaques with visual diameter stenosis >20% on CCTA
5. At the baseline visit, participants must be on a stable (>4 weeks) regiment of diabetes medications.
6. Patients using oral hormonal contraceptives must switch to a non-oral contraceptive method, or add a barrier method of contraception for 4 weeks after initiation and for 4 weeks after each dose escalation

Exclusion Criteria:

1. Have had a major cardiovascular event within the last 60 days
2. Have type 1 diabetes mellitus
3. Current use of GLP1-RA
4. Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the last 6 months
5. Are currently planning treatment for diabetic retinopathy and/or macular edema
6. Have history of, or currently planning a coronary, carotid, or peripheral artery revascularization (ie - stent, bypass)
7. Have a history of pancreatitis
8. Have a history of ketoacidosis or hyperosmolar state/coma
9. Have a known clinically significant gastric emptying abnormality, have undergone or currently planning any gastric outlet obstruction, or have undergone or currently planning any gastric bypass (bariatric) surgery or restrictive bariatric surgery
10. Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years
11. Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
12. Have had a blood transfusion or severe blood loss within 90 days prior to screening or have known hematological conditions that may interfere with HbA1c measurement
13. Planned or Prior Bypass surgery
14. Contradiction for CCTA (e.g. serious allergic reaction to the contrast dye) or CCTA not meeting entry standards after two attempts during the Baseline CCTA visit as assessed by the imaging core lab.
15. Uncontrolled severe hypertension: systolic blood pressure > 180 mmHg or diastolic BP > 100 mm Hg prior to randomization (assessed at the screening visit) despite antihypertensive therapy
16. Heart Failure NYHA Class III or IV at the screening visit
17. Renal insufficiency (eGFR <40 ml/min/1.73m2) as measured by the Modification of Diet in Renal Disease (MDRD) formula at the screening visit.
18. Hospitalization for major cardiovascular event including heart failure in the past 2 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of total non-calcified coronary plaque volume | 12 months
  Reduction of total non-calcified coronary plaque volume from baseline (start of the study) till the final visit will be measured using Coronary Computed Tomography Angiography (CCTA).

SECONDARY OUTCOMES:
Reduction of low attenuation plaque volume | 12 months
  Reduction change in low attenuation plaque volume from baseline (start of the study) till the final visit will be measured using Coronary Computed Tomography Angiography (CCTA)
Reduction of total plaque volume, fibrous, lipid-rich and calcified plaque volumes using CCTA | 12 months
  Reduction change of total plaque volume, fibrous, lipid-rich and calcified plaque volumes will be compared between baseline and at the end of the study.
Change in HgA1c lab values in the blood. | 12 months
  Change in HgA1c lab values in the blood will be compared between baseline and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Budoff, MD, Principal Investigator — The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center (The Lundquist Institute), Torrance, California, United States